CLINICAL TRIAL: NCT03777488
Title: Pharmacokinetics of Tranexamic Acid After Oral, Intramuscular or Intravenous Administration: a Prospective, Randomised, Cross-over Trial in Healthy Volunteers.
Acronym: PharmacoTXA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/KEP/205
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteer Study
Keywords: pharmacokinetics, tranexamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Tranexamic acid Group 1 (Experimental): Participants will receive tranexamic acid in the following order:
  First Dose: Intravenous Second Dose: Intramuscular Third Dose: Oral
  Interventions: Drug: Tranexamic Acid 1 gram intravenously; Drug: Tranexamic acid 2 grams oral solution; Drug: Tranexamic acid 1 gram intramuscular
- Tranexamic acid Group 2 (Experimental): Participants will receive tranexamic acid in the following order:
  First Dose: Intravenous Second Dose: Oral Third Dose: Intramuscular
  Interventions: Drug: Tranexamic Acid 1 gram intravenously; Drug: Tranexamic acid 2 grams oral solution; Drug: Tranexamic acid 1 gram intramuscular
- Tranexamic acid Group 3 (Experimental): Participants will receive tranexamic acid in the following order:
  First Dose: Intramuscular Second Dose: Intravenous Third Dose: Oral
  Interventions: Drug: Tranexamic Acid 1 gram intravenously; Drug: Tranexamic acid 2 grams oral solution; Drug: Tranexamic acid 1 gram intramuscular
- Tranexamic acid Group 4 (Experimental): Participants will receive tranexamic acid in the following order:
  First Dose: Intramuscular Second Dose: Oral Third Dose: Intravenous
  Interventions: Drug: Tranexamic Acid 1 gram intravenously; Drug: Tranexamic acid 2 grams oral solution; Drug: Tranexamic acid 1 gram intramuscular
- Tranexamic acid Group 5 (Experimental): Participants will receive tranexamic acid in the following order:
  First Dose: Oral Second Dose: Intravenous Third Dose: Intramuscular
  Interventions: Drug: Tranexamic Acid 1 gram intravenously; Drug: Tranexamic acid 2 grams oral solution; Drug: Tranexamic acid 1 gram intramuscular
- Tranexamic acid Group 6 (Experimental): Participants will receive tranexamic acid in the following order:
  First Dose: Oral Second Dose: Intramuscular Third Dose: Intravenous
  Interventions: Drug: Tranexamic Acid 1 gram intravenously; Drug: Tranexamic acid 2 grams oral solution; Drug: Tranexamic acid 1 gram intramuscular

INTERVENTIONS:
Drug: Tranexamic Acid 1 gram intravenously — Intravenous tranexamic acid crossover to oral and intramuscular arms
Drug: Tranexamic acid 2 grams oral solution — Oral tranexamic acid crossover to intravenous and intramuscular arms
Drug: Tranexamic acid 1 gram intramuscular — Intramuscular tranexamic acid crossover to oral and intravenous arms

SUMMARY:
This is a Phase 1 study which aims to determine the pharmacokinetics and local and systemic tolerance of tranexamic acid in healthy volunteers using a population approach after oral, intramuscular or intravenous administration. It will also determine the feasibility of measuring tranexamic acid in spots of dry capillary blood.

DETAILED DESCRIPTION:
Fifteen healthy volunteers will receive in random order 1 gram of intravenous and intramuscular injections and 2 grams of oral tranexamic acid solution. Blood samples will be taken at:

* T0+ 5min (only for IV route)
* T0+30min
* T0+1h
* T0+2h
* T0+3h
* T0+4h
* T0+5h
* T0+6h
* T0+8h (only for IM and PO routes)
* T0+24h

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers both men and non-pregnant women
* ≥18-≤45-year-old
* Body mass index between ≥18 and ≤30 kg/m2, and bodyweight between ≥50 and ≤100 kg
* Coagulation test results of fibrinogen, D-dimers, prothrombin time and a partial thromboplastin time within normal limits at screening
* Normal renal function based on medical history and laboratory tests
* If a woman, must have a negative urine β-human chorionic gonadotropin (βhCG) pregnancy test at screening and inclusion visits
* Provision of signed informed consent prior to any study specific procedure
* People with public healthcare insurance (in France)

Exclusion Criteria:

* Previous thrombotic event or pre-existing pro-thrombotic disease
* Any history of seizures
* Any chronic or active cardiovascular or renal disease
* Planned general anaesthesia or surgery in the 3 months following inclusion
* Pregnant and/or breastfeeding
* Known allergy to the study drugs or any of the excipients of the formulations
* Use of any prescription or non-prescription medication (other than hormonal contraception) within 7 days before the first dose of the study drug is scheduled
* Inability to give informed consent
* Previous participation during the year in clinical studies compensated for an amount incompatible with participation in this study, verified by recording in the national register of subjects participating in human research trials
* Legal criteria:

  * People deprived of liberty by judicial or administrative decision
  * Adult protected by law (France)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Serum tranexamic acid concentrations versus time profiles for each route of administration (Oral, intramuscular and intravenous) | 24 hours

SECONDARY OUTCOMES:
Pain during after administration (visual analogue scale) for each administration route | 8 hours
  (Scale 0 - 9) where 0 = no pain and 9 most severe pain
Reaction at site of injection for intramuscular and Iintravenous routes | 24 hours
• Correlation between serum and dry blood spot concentrations for each administration route | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Haleema Shakur-Still, Study Chair — London School of Hygiene and Tropical Medicine; Ian Roberts, Study Chair — London School of Hygiene and Tropical Medicine
Locations (2):
- France (2):
  - UFR Sciences de la Santé Simone Veil Université Versailles Saint Quentin en Yvelines, Montigny-le-Bretonneux
  - Unité de Recherche Clinique Paris Descartes Necker Cochin, Hôpital Necker-Enfants Malades, Paris

REFERENCES:
- [Derived] Grassin-Delyle S, Semeraro M, Lamy E, Urien S, Runge I, Foissac F, Bouazza N, Treluyer JM, Arribas M, Roberts I, Shakur-Still H. Pharmacokinetics of tranexamic acid after intravenous, intramuscular, and oral routes: a prospective, randomised, crossover trial in healthy volunteers. Br J Anaesth. 2022 Mar;128(3):465-472. doi: 10.1016/j.bja.2021.10.054. Epub 2022 Jan 5. PMID 34998508